CLINICAL TRIAL: NCT02032979
Title: Neurological and Psychiatric Comorbidities Patients With FSHD 1 and 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-AOI-06
Record Dates: First submitted 2013-12-10; First posted 2014-01-10 (Estimated); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Muscular Dystrophy, Facioscapulohumeral
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FSHD patient (Experimental)
  Interventions: Behavioral: Psychiatric test

INTERVENTIONS:
Behavioral: Psychiatric test

SUMMARY:
The investigators propose to conduct a comparative pilot cognitive and psychiatric profiles of 10 patients Facio-Scapulo-Humeral Dystrophy (= FHSD) type 1 and 10 patients with type 2 FSHD study. For this, the investigators relied on observational components: FSHD2 patients appear more often present with psychiatric comorbidities and seem to have lower cognitive performance compared to FSHD1 patients. This was confirmed by a preliminary study on a small sample population of patients. It seems to exist mainly executive dysfunction associated with attention disorders in patients FSHD2. Moreover, their performance in IQ tests would be low in relation to their socio-educational and compared with patients FSHD1 level.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years and <75 years
* FSHD patients 1 or 2 with genetic confirmation

Exclusion Criteria:

* Phosphokinase creatine level > 5 time of the normal
* Patient as medical history :

  * A history or active neurological disease likely to interfere with the interpretation of results
  * a history of head trauma
  * an infectious disease, hormonal, inflammatory or some deficiency may induce cognitive and / or psychiatric troubles
  * Patient with cons-indication for performing a brain MRI
* Pregnant, parturient and lactating (producing a serum pregnancy test)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-10-20 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Montgomery and Asberg Depression Rating Scale | One time at the inclusion
Hamilton Depression Rating Scale | One time at the inclusion
Hamilton Anxiety Rating Scale | One time at the inclusion
Quick inventory of depressive symptomatology Self report | One time at the inclusion
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form | One time at the inclusion
Mini Mental Status Evaluation | One time at the inclusion
Wechsler Adult Intelligence Scale | One time at the inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pasteur, Nice, France